CLINICAL TRIAL: NCT03198156
Title: Transcranial Direct Current Stimulation Therapy for Central Hypersomnia Without Cataplexy
Acronym: tDCS
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Funding Stopped
Sponsor: Ohio State University (Other)
Collaborators: United States Air Force (U.S. Federal Agency)
Responsible Party: Principal Investigator, Ulysses Magalang MD, Professor of Medicine and Neuroscience; Director, Sleep Medicine Program, Ohio State University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2016H0434
Record Dates: First submitted 2017-06-21; First posted 2017-06-26 (Actual); Results first posted 2021-10-25 (Actual); Last update posted 2021-10-25 (Actual); Status verified 2021-10

CONDITIONS: Hypersomnia
Keywords: Transcranial Direct Current Stimulation; Without Cataplexy
MeSH Terms: conditions — Disorders of Excessive Somnolence | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Intervention Model Description: This is a 5 week randomized, sham-controlled, parallel group study involving subjects with any of the following diagnoses: Idiopathic Hypersomnia, Narcolepsy without Cataplexy, Hypersomnia in OSA patients adequately treated with PAP therapy or dental device, Posttraumatic hypersomnia, Hypersomnia, unspecified. Subjects with idiopathic hypersomnia with an MSLT mean sleep latency of >8 minutes will undergo actigraphy and those with an average sleep time of >10 hours per day will continue with the study while those with <10 hours sleep time will be excluded. OSA subjects with complaints of hypersomnia with an ESS score <10 will be excluded. Female subjects of child bearing age and not menopausal will have a pregnancy test performed.
  Subjects will receive either active tDCS or sham stimulation for 30 minutes daily for 4 sessions. Subjects will be blinded as to whether they are receiving sham or active tDCS treatments.
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Transcranial Direct Current Stimulation (Experimental): Active tDCS for 30 minutes daily for 4 sessions
  Interventions: Device: Transcranial Direct Current Stimulation
- Sham stimulation (Sham Comparator): Sham stimulation sessions will be for 30 minutes daily for each of the 4 sessions; however, active stimulation for this arm of the study is only for 30 seconds; yet, will be applied at the same intensity as the Active arm of the study, albeit for only 30 seconds.
  Interventions: Device: Sham stimulation

INTERVENTIONS:
Device: Transcranial Direct Current Stimulation — tDCS is a form of noninvasive, painless, brain stimulation that uses a mild direct electrical current passed between electrodes on the scalp to modify neuronal membrane resting potential in a polarity dependent manner, elevating or lowering neuron excitability in a region.
  Other Names: tDCS
  Arms: Transcranial Direct Current Stimulation
Device: Sham stimulation — Sham stimulation
  Arms: Sham stimulation

SUMMARY:
1. To determine the effects of transcranial direct current stimulation (tDCS) on vigilance in subjects with central hypersomnia without cataplexy.
2. To determine the effects of tDCS on subjective measures of sleepiness and alertness in subjects with central hypersomnia without cataplexy.

DETAILED DESCRIPTION:
This is a randomized, sham-controlled, parallel group study. The study will last up to 5 weeks. After informed consent, subjects with idiopathic hypersomnia with an MSLT mean sleep latency of >8 minutes will undergo actigraphy and those with an average sleep time of >10 hours per day will continue with the study while those with <10 hours sleep time will be excluded. In addition, OSA subjects with complaints of hypersomnia with an ESS score <10 will also be excluded. Female subjects of child bearing age and not menopausal will have a pregnancy test performed as pregnancy is an exclusionary criteria.

Subjects will be randomized to receive either active tDCS or sham stimulation for 30 minutes daily for 4 sessions. The randomization will be generated by means of a computer-generated random-number table. An unrestricted randomization scheme will be followed. Subjects will be blinded as to whether they are receiving sham or active tDCS treatments. The investigator who will conduct the analysis of all outcomes will be blinded as to subject treatment assignment.

All stimulation visits will be completed within a five-consecutive day period; that is one stimulation visit may be missed provided a total of four stimulation visits are completed within a five-day period. Outcome measures will include: psychomotor vigilance test (PVT), subjective measures of sleepiness, and the Center for Epidemiologic Studies Depression (CES-D) scale. PVT will be performed pre- and post- stimulation during the first and last stimulation sessions. Subjective measures of sleepiness include the following: Epworth Sleepiness Scale (ESS), Stanford Sleepiness Scale (SSS), Functional Outcomes of Sleep Questionnaire-10 (FOSQ-10), and Visual Analogue Scale (VAS).

ELIGIBILITY:
Inclusion Criteria:

* Age 18 - 70 years
* Epworth Sleepiness scale score >10
* Stable medication dosage over previous 4 weeks
* Able to understand English and read and write at the 8th grade level and give a written informed consent document.
* Stable sleep/wake schedule (that is, no rotating shift work)
* Clinical diagnosis of any of the following:

  1. Idiopathic Hypersomnia
  2. Narcolepsy without Cataplexy
  3. Hypersomnia in OSA patients adequately treated with PAP therapy or dental device
  4. Posttraumatic hypersomnia
  5. Hypersomnia, unspecified
* Multiple sleep latency test (MSLT) shows fewer than two sleep onset REM periods and a mean sleep latency of ≤ 8 minutes. An MSLT is not required for inclusion of OSA patients provided their Epworth Sleepiness Scale (ESS) score is >10. Adequately treated OSA patients will be defined as: i) an average PAP usage of > 4 hours per night and a residual apnea-hypopnea index (AHI) of <10/hour based on PAP machine download during at least a 30-day period, or ii) regular use of dental device during sleep based on self-report and a prior sleep study showing an AHI <10/hour while using the dental device.
* Subjects with idiopathic hypersomnia with an MSLT mean sleep latency of > 8 minutes will be included provided they have hypersomnia symptoms and habitually long sleep times (average of >10 hours per day) documented by actigraphy for at least 7 days.18

Exclusion Criteria:

* Self-reported habitual sleep period of < 7 hours/night
* History of automobile accident due to falling asleep while driving
* Currently taking stimulant medications such as Modafinil, Armodafinil, Methylphenidate, or Dextroamphetamnie.
* Inability to understand or read English
* Clear history of cataplexy
* Moderate or severe sleep apnea defined as an apnea-hypopnea index (AHI) of > 15/hour based on a previous sleep study and non-compliant with treatment.
* Self-reported Substance abuse (current)
* Excessive alcohol consumption defined as:
* More than 3 glasses of wine a day
* More than 3 beers a day
* More than 60 mL of hard liquor a day
* Presence of cardiac pacemaker or automatic implantable cardioverter-defibrillator (AICD).
* Pregnancy, lactation
* Recent hospitalization for major surgery/major illness (within past 1 month)
* Non-removable metal or tattoos around head
* Use of implantable birth control device such as Implanon
* History of severe and frequent headaches
* Known coronary artery disease
* Seizure disorder
* Uncontrolled hypertension
* Congestive heart failure

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2017-09-01 (Actual); Primary Completion 2020-06-20 (Actual); Study Completion 2020-06-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ulysses Magalang, MD, Principal Investigator — Ohio State University
Locations (1):
- The Ohio State University, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Of 39 enrolled subjects, 38 met inclusion criteria and were randomized to treatment
Period: Overall Study
Arm/Group | Transcranial Direct Current Stimulation | Sham Stimulation
Started | 19 | 19
Completed | 19 | 19
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Transcranial Direct Current Stimulation | Sham Stimulation | Total
Number analyzed (Participants) | 19 | 19 | 38
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: A total of 38 subjects age data were analyzed
  years | 38.63 (11.34) | 38.84 (14.27) | 38.73 (25.61)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 12 | 22
  Male | 9 | 7 | 16
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 3 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 1 | 3
  White | 15 | 15 | 30
  More than one race | 2 | 0 | 2
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 19 | 19 | 38
BMI [Mean (Standard Deviation); unit: kg/m^2] — Population: A total of 38 subjects BMI were analyzed
  kg/m^2 | 29.70 (5.02) | 29.84 (6.67) | 29.77 (5.26)

OUTCOME MEASURES:

1. Primary Outcome: Psychomotor Vigilance Test
Description: Objective measure of sleepiness.
Time Frame: 10 minutes
Population: Sleepiness measure data based on Psychomotor Vigilance Test results could not be analyzed and reported in the table data as we were unable to collect data from enrolled patients.
Arm/Group | Transcranial Direct Current Stimulation | Sham Stimulation
Number analyzed (Participants) | 0 | 0

2. Primary Outcome: Epworth Sleepiness Scale
Description: Subjective measure of sleepiness
Time Frame: 5 minutes
Population: Subjective Sleepiness data based on patient report on the Epwoth Sleepiness Scale questionnaire could not be analyzed and reported in data table as were unable to be collect data from enrolled patients. This study terminated early.
Arm/Group | Transcranial Direct Current Stimulation | Sham Stimulation
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Stanford Sleepiness Scale
Description: Subjective measure of sleepiness
Time Frame: 5 minutes
Population: Subjective Sleepiness data based on Stanford Sleepiness Scale instrument could not be analyzed and reported in the table data as we were unable to collect data from enrolled patients. This study was early terminated.
Arm/Group | Transcranial Direct Current Stimulation | Sham Stimulation
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Functional Outcomes of Sleep Questionnaire
Description: Measure of the impact of sleepiness on daytime function
Time Frame: 5 minutes
Population: Impact of sleepiness on daytime function based on functional outcomes of sleep questionnaire could not be analyzed and reported in the table data as we were unable to collect data from enrolled patients.
Arm/Group | Transcranial Direct Current Stimulation | Sham Stimulation
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Visual Analogue Scale
Description: Subjective Measure of Sleepiness
Time Frame: 5 minutes
Population: Subjective Sleepiness data based on Visual Analogue Scale (VAS) could not be analyzed and reported in the table data as we were unable to collect data from enrolled patients.
Arm/Group | Transcranial Direct Current Stimulation | Sham Stimulation
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: CES-D Scale
Description: Center for Epidemiologic Studies Depression (CES-D) Scale
Time Frame: 5 minutes
Population: Data from Center for Epidemiologic Studies Depression (CES-D) Scale could not be analyzed and reported in the table data as we were unable to collect data from enrolled patients
Arm/Group | Transcranial Direct Current Stimulation | Sham Stimulation
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse events were assessed through study completion (5 weeks for each participant).
Description: No adverse events were observed or reported during the study.
Arm/Group | Transcranial Direct Current Stimulation | Sham Stimulation
All-Cause Mortality (participants affected / at risk) | 0/19 | 0/19
Serious Adverse Events (participants affected / at risk) | 0/19 | 0/19
Other Adverse Events (participants affected / at risk) | 0/19 | 0/19

LIMITATIONS AND CAVEATS:
No data was analyzed. Study was terminated due to the funding was stopped.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-05-29): https://cdn.clinicaltrials.gov/large-docs/56/NCT03198156/Prot_SAP_002.pdf
  • Informed Consent Form (2020-01-17): https://cdn.clinicaltrials.gov/large-docs/56/NCT03198156/ICF_003.pdf